CLINICAL TRIAL: NCT05619458
Title: Effectiveness of an Adapted Version of the Learning to BREATHE Program on Emotion Regulation Among Youth Attending an Alternative High School: Rationale and Design for a Single-arm Trial
Brief Title: Effectiveness of a Mindfulness Program on Emotion Regulation Among Youth Attending an Alternative School
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lethbridge (Other)
Responsible Party: Principal Investigator, Cheryl Currie, Associate Professor, University of Lethbridge
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ULethbridge
Record Dates: First submitted 2022-11-08; First posted 2022-11-16 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Substance Use; Mindfulness; Adolescent Behavior; Emotion Regulation; Social Behavior; Self Esteem
MeSH Terms: conditions — Substance-Related Disorders; Adolescent Behavior; Emotional Regulation; Social Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness intervention (Experimental): The intervention will consist of 6 one-hour sessions delivered once per week in a classroom at an alternative high school during normal school hours.
  Interventions: Behavioral: Mindfulness Intervention

INTERVENTIONS:
Behavioral: Mindfulness Intervention — 6-week mindfulness intervention
  Other Names: Learning to Breathe Program

SUMMARY:
The main goal of this single-arm pre-post intervention study is to see if an adapted mindfulness program can improve emotion regulation among youth aged 15-19 years who attend an alternative school. Participants will complete a baseline survey package using an iPad. They will then receive an adapted version of the 6-session Learning to BREATHE Program as part of a course they are taking at their school. Students will again complete a survey package within 2 weeks of completing the program. The investigator will compare baseline and post-intervention survey responses to see if the program improved emotion regulation, as well as several secondary psychosocial and behavioral outcomes.

DETAILED DESCRIPTION:
BACKGROUND: The purpose of this study is to use a single-arm trial to assess the effectiveness of a 6-week mindfulness-based intervention (MBI) on the emotional, social, and behavioural well-being of adolescents attending an alternative school in Lethbridge, Alberta. Mindfulness focuses on cultivating present-moment awareness in a non-reactive and non-judgmental way. A 2017 meta-analysis found MBIs have a moderate effect on increasing mindfulness among youth in controlled studies. A 2020 meta-analysis found MBIs have an overall small effect size over a broad range of samples and mental health outcomes among youth. The review found that in clinical samples of youth the effect size for mental health outcomes is in the moderate range, and nearly three times the magnitude found of non-clinical samples. MBIs also improve the mental health of at-risk youth including those in foster care, prison, and those who are survivors of interpersonal trauma. The goal of the present study is to build upon emerging evidence suggesting MBIs may be a useful addition to the curriculum within an alternative school environment. Alternative schools, also called outreach schools in Alberta, address the interpersonal, social, and learning needs of teens that cannot be met in regular school settings. Alternative schools offer a flexible learning environment with innovative programming designed to provide academic, social and emotional supports and skill building. Youth who attend alternative schools experience more psychosocial problems, including adverse childhood experiences (ACEs), and health risk behaviours; and thus may benefits from MBIs. Learning how to regulate emotions in a socially adaptive and appropriate manner is an important part of healthy psychological development. Emotion regulation allows an adolescent greater autonomy, strengthens self-esteem and improves self-efficacy. The poor regulation of emotions is implicated in the diagnostic criteria of many mental health disorders. It is generally agreed in the literature that emotion regulation processes can be conscious or unconscious, and automatic or effortful. It is also generally agreed that emotion regulation involves both reducing the intensity and frequency of negative emotional states, as well as developing the ability to create and maintain positive emotions. While MBIs have been shown to strengthen emotion regulation in regular public high schools, the extent to which MBIs strengthen emotion regulation within alternative schools is not well understood, and the primary focus of the present study. The investigator will also explore the impact of an MBI intervention on mindfulness, psychological outcomes, social connection, and behaviour.

INTERVENTION: In this study, the investigator will use the six-week, evidence-based Learning to BREATHE Program as the primary intervention. Learning to BREATHE teaches emotion regulation and stress-reduction in relatable ways for teens. The program is delivered flexibly and adaptively rather than as a manualized curriculum, which fits the learning environment and goals of alternative schools. To date, two studies have examined the effectiveness of the Learning to BREATHE program in alternative schools. The first study, based in the US, used a pre-post design and found significant improvements in self-esteem and perceived stress. The second study used a randomized controlled design with an active comparator to assess Learning to BREATHE against a program designed to reduce substance use. The team reported many intervention delivery problems within an alternative school, including youth who were disinterested and disruptive during sessions. Changes were made to the intervention throughout the trial to address these problems, including involving teachers and school support staff in the sessions as youth were more familiar and comfortable with them. They also shortened activities that youth found difficult (sitting meditation), and lengthening others that youth enjoyed (body scan meditations and restorative yoga exercises). At study end, the Learning to BREATHE program intervention was more effective at reducing depression than active control. However, the small sample size (N = 14 intervention, N = 13 active control) and changes to the intervention throughout the trial made it difficult to assess impacts. To address these problems before the present study began, the investigator worked with social workers, school administrators, and community stakeholders in 2018-2019 to adapt the Learning to BREATHE Program for delivery within an alternative school environment. Suggested adaptions for program delivery were pilot tested in 2019-20 in a small sample of junior high students (N = 17) in the Lethbridge Alternative School Program. Sessions were delivered by three facilitators with mindfulness training certification. Due to the COVID-19 pandemic intervention effectiveness could not be assessed. The investigator was limited to analyzing post-intervention data collected before government-mandated school closures in March 2020 (N = 6 of 17 students who took part in the program). Fidelity and observational data collected during each session was also analyzed, and used in a student MSc thesis. The findings suggest youth were engaged in the adapted version of the program, that their understanding of mindfulness as a tool for stress and coping increased, and that incorporating digital technology (apps) to deliver segments of the intervention promoted independent use of the digital tools by youth outside the sessions.

METHODS: This intervention study will begin November 28, 2022, at a single location - Victoria Park High School in Lethbridge, AB. The study will be led by Dr. Cheryl Currie in the Faculty of Health Sciences at the University of Alberta in Alberta, Canada. The study is expected to end January 31, 2023. It is estimated that from time of first contact during student enrolment in the study each participant will be engaged in the study for nine weeks, excluding time away during the December holiday break. This includes one week to complete the pre-intervention data collection meeting with school staff, six weeks to take part in the intervention, and up to two weeks to complete a post-intervention data collection meeting with a school staff member. This study will recruit a school-based sample of approximately 35 youth that meet eligibility criteria to achieve 31 participants. Participants will be students registered in two specific classes in Victoria Park High School. These courses were chosen by school administration for participation in the program. A low (5%) loss to follow-up is expected given the program will be offered as part of two combined courses that students have chosen to enroll in. Students will complete the baseline survey immediately after completing the informed consent process by clicking the second Qualtrics tab that will be open on their iPad browser. The survey will be administered using the Qualtrics survey platform on iPads provided by the University of Lethbridge study team and will take approximately 20 minutes. Within two weeks of completing the intervention, participants will complete the same survey package they answered at baseline.

ANALYSIS STRATEGY: Data will be analyzed using Stata 17.0 and R software. The investigator will use frequencies and percentages to summarize participant age, grade, genders, Indigenous status (identify as Indigenous - yes or no), immigrant status (born in Canada - yes or no), and who participants currently live with. The purpose of collecting this data is to create a broad, general description of the sample in dissemination documents. For prediction of emotion regulation pre- and post-intervention, participants will be included in the analysis if they have completed 50% of the intervention and completed follow-up data collection. Missing data for participants who meet these criteria will be addressed using multiple imputation. A repeated-measures, mixed-model approach will be used to identify significant changes in each of the primary and secondary outcomes pre-post intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged 15-19 years of age
* Enrolled in two specific courses offered at Victoria Park High School

Exclusion Criteria:

* Unwilling to give consent
* Lack capacity to provide informed consent as determined by the educational assistant who will complete the informed consent process with each potential participant.

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline in emotion regulation on the 18-item Difficulties in Emotion Regulation Scale - Short Form (DERS-SF) | Baseline and Week 10
  The DERS-SF has excellent psychometric properties regardless of age and gender variation. A 5-point Likert scale from 1 (almost never) to 5 (almost always) is employed, with higher scores indicating greater emotion regulation impairment or dysregulation (Week 10 Score - Baseline Score)
Change from baseline in emotion regulation on the 1-item Emotion Regulation Questionnaire for Children and Adolescents (ERQ-CA) | Baseline and Week 10
  The ERQ-CA assesses use of two emotion regulation strategies: cognitive reappraisal where a person attempts to change how they think about a situation to change its emotional impact, and expressive suppression where a person attempts to inhibit the behavioural expression of their emotions. A 5-point Likert scale from 1 (almost never) to 5 (almost always) is employed, with higher scores indicating greater emotion regulation impairment or dysregulation (Week 10 Score - Baseline Score).

SECONDARY OUTCOMES:
Change from baseline in mindfulness on the 10-item Child and Adolescent Mindfulness Measure (CAMM). | Baseline and Week 10
  The CAMM has good internal reliability in a variety of adolescent populations, with Cronbach's alpha scores reported between 0.80-0.84, and no significant gender differences. The measure uses a 5-point Likert scale with higher scores indicated greater mindfulness (Week 10 Score - Baseline Score).
Change from baseline in anxiety and depression symptoms on the 4-item Patient Health Questionnaire (PHQ-4). | Baseline and Week 10
  The PHQ-4 is a reliable measure of anxiety (α = 0.82) and depression (α = 0.81) separately and in composite (α = 0.85). Items are measured on a 4-point Likert scale, with options ranging from "Not at all" to "Nearly every day", with higher scores indicating more frequent anxiety/depression symptoms (Week 10 Score - Baseline Score).
Change from baseline in self-esteem on the 5-item Brief Rosenberg Self-Esteem Scale. | Baseline and Week 10
  The Brief Rosenberg Self-Esteem Scale assesses self-esteem by asking participants to reflect on the feelings they have about themselves using a 4-point scale ranging from strongly agree to strongly disagree, with higher scores indicating higher self-esteem (Week 10 Score - Baseline Score).
Change from baseline in school connectedness on an adapted version of the the National Longitudinal Study of Adolescent Health School Connectedness Scale (NLSAH-SCS). | Baseline and Week 10
  The version of the NLSAH-SCS that will be used in this study was developed by investigators of the COMPASS Study - a prospective cohort study that collects longitudinal data from a sample of grade 9-12 in Canada. The adapted measure predicts reduced health risk behaviour in Canadian high school students. Consistent with the original measure, response options range from 1=strongly disagree to 4=strongly agree, with higher scores indicating stronger feelings of school connectedness (Week 10 Score - Baseline Score).
Change from baseline in home connectedness on an adapted 5-item version of the National Longitudinal Study of Adolescent Health School Connectedness Scale (NLSAH-SCS). | Baseline and Week 10
  We have adapted the 5-item measure of school connectedness to measure an adolescent's sense of connectedness within their home (e.g., I feel close to people in my home, I feel safe in my home, I feel the adults in my home treat me fairly). Consistent with the original measure, response options range from 1=strongly disagree to 4=strongly agree, with higher scores indicating stronger feelings of connectedness at home (Week 10 Score - Baseline Score).
Change from baseline in substance use on the Screen for Substance-Related Risks and Problems in Adolescents (CRAFFT) 2.1+N | Baseline and Week 10
  CRAFFT scores are strongly correlated with diagnostic classifications for substance use among adolescents. We will use the new 2.1+N version of the CRAFFT which also assess tobacco use and vaping. All questions have yes/no responses, with higher scores indicating more significant substance use and problems (Week 10 Score - Baseline Score).

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Currie, PhD, Principal Investigator — University of Lethbridge
Locations (1):
- Victoria Park High School, Lethbridge, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No